CLINICAL TRIAL: NCT06246890
Title: Autism Access Link for Early Referral and Treatment Expansion
Brief Title: Autism ALERT Expansion
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00020673
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Primary Care; Case Management
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics; Caffeine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening + Autism ALERT: Families with children under 54 months, without a medical ASD diagnosis, who are referred by an autism clinic or primary care provider to Autism ALERT
  Interventions: Other: Autism ALERT

INTERVENTIONS:
Other: Autism ALERT — Autism Access Link for Early Referral and Treatment [ALERT], the intervention proposed in this application, is a novel state-wide referral and case management platform that PCPs can activate to ensure that a child with suspected ASD receives all necessary ASD diagnosis and treatment resources in a single referral, radically simplifying a complex diagnostic and treatment process.
  Other Names: Autism Access Link for Early Referral and Treatment [ALERT]

SUMMARY:
Autism Access Link for Early Referral and Treatment [ALERT], the intervention proposed in this application, is a novel state-wide referral and case management platform that PCPs can activate to ensure that a child with suspected ASD receives all necessary ASD diagnosis and treatment resources in a single referral, radically simplifying a complex diagnostic and treatment process. We hypothesize that Autism ALERT will have strong acceptability and high rates of use among primary care providers as well as among diverse low-income parents of children at risk for ASD, and that we will see increased rate of child ASD educational evaluations within six months, and shortened time between referral and ASD treatment.

DETAILED DESCRIPTION:
Though significant research effort has focused on autism spectrum disorder (ASD) screening, less attention has been devoted to optimizing follow-up of children who are subsequently identified as at-risk. Despite increases in ASD screening rates, many children with ASD wait years between when autism is suspected in the primary care setting and when definitive diagnosis and treatment begin. Delayed and missed diagnoses are particularly problematic for low-income and racial/ethnic minority children in the US, who experience higher rates of these adverse outcomes.

The Autism Access Link to Early Referral and Treatment (Autism ALERT) program is a statewide monitoring and case management program to accelerate access to ASD diagnosis and treatment among children with suspected ASD the primary care setting. The system will reduce the time between identification of suspected ASD in the primary care setting and establishment of ASD diagnosis and treatment services, by reducing family barriers to care, decreasing primary care provider burdens, and simplifying referral processes. Following an initial pilot trial, we propose implementing the intervention to families in the Portland metropolitan area before expanding the program elsewhere in the state. The program will be available to any Oregon child age 12-54 months, regardless of health system or payor type. Autism ALERT will become part of the Help Me Grow national network, which gives it potential for statewide and national spread.

In this proposed research, we will undertake a single arm implementation/effectiveness trial in which the program will be tested throughout the state of Oregon, beginning in the Portland metropolitan area. In the long term, this research will result in a sustainable, evidence-based statewide and ultimately national monitoring system children with suspected ASD.

ELIGIBILITY:
Inclusion Criteria:

* child's primary care provider suspects the child has ASD
* child is a patient at one of the study clinics
* child age 12 to 54 months
* family speaks English or Spanish
* no prior ASD medical diagnosis or ASD diagnostic evaluation

Exclusion Criteria:

- Previous diagnosis of ASD or prior diagnostic evaluation for ASD.

Ages: 12 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Families with a child aged 12-54 months who are suspected to have autism by a primary care provider who have not received a medical autism diagnosis or a prior diagnostic autism evaluation. Initially restricted to residents of the Multnomah, Clackamas, or Washington counties of Oregon.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in satisfaction with Care Coordination in general and for autism in particular | At enrollment and study end (~9 months after enrollment)
  2 separate provider survey measures
Change in Parent stress | At enrollment and 6 months after enrollment
  Parent Survey - Parenting Stress Index
Change in Parenting stress | At enrollment and 6 months after enrollment
  Questionnaire on Resources and stress - Short Form
Change in Family Empowerment | At enrollment and 6 months after enrollment
  Parent Survey - Family Empowerment Scale, Family Subscale
Change in Family Centered and Coordinated Care | At enrollment and 6 months after enrollment
  Parent Survey - Items from National Survey of Children's Health, Medical Home item set
Family Satisfaction with Program | 6 months after enrollment
  Parent Survey items - Satisfaction with Interpersonal Relationship with Navigator (PSN-I), Client Satisfaction Questionnaire - 8
% referred to program who complete an ASD educational evaluation within 6 months | 6 months after enrollment
  Administrative data - Oregon Early Intervention/Early Childhood Special Ed (EI/ECSE) database
Time from EI/ECSE referral to ASD treatment in EI/ECSE, among children with ASD | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
Family self-reported ASD knowledge | At enrollment and 9 months after enrollment
  5-item survey measure
Change in provider self-efficacy about autism management | At enrollment and at study end (~9 months after enrollment)
  1-item survey measure

SECONDARY OUTCOMES:
Change in provider autism paperwork burden | At enrollment and at study end (~9 months after enrollment)
  Provider survey item
Time from EI/ECSE referral to evaluation among children with ASD | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
Age of EI/ECSE educational determination, among children with ASD | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
% with ASD determination receiving ASD services 6 months after enrollment | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
monthly service hours among children with ASD 6 months after enrollment | measured 9 months after enrollment
  Administrative data - Oregon EI/ECSE database
age of ASD medical diagnosis among children on Medicaid | Measured 1 year after study enrollment
  Administrative data - Medicaid claims
% with ASD medical diagnosis receiving ASD therapy 6 months after enrollment, among children on Medicaid | Measured 1 year after study enrollment
  Administrative data - Medicaid claims

CONTACTS AND LOCATIONS:
Locations (1):
- Ohsu Cdrc, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT06246890/Prot_000.pdf